CLINICAL TRIAL: NCT00700518
Title: A Phase I Trial of the Pharmacodynamic Dose Response to Topical Trinitrate in Patients With Raynaud's Phenomenon
Brief Title: Dose Response to Topical Glyceryl Trinitrate in Patients With Raynaud's Phenomenon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procris Pharmaceuticals (Industry)
Responsible Party: Matthew A. Gonda, Ph.D, Procris Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150-005
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Raynaud's Phenomenon
Keywords: Raynaud's Syndrome; Raynaud's Disease; RP
MeSH Terms: conditions — Raynaud Disease | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1. (Placebo Comparator): placebo cream applied to 2 adjacent fingers on non-dominant hand one time
  Interventions: Drug: placebo cream
- 2 (Active Comparator): 0.6mg of Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand
  Interventions: Drug: Glyceryl Trinitrate
- 3 (Active Comparator): 1.2mg of Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand one time
  Interventions: Drug: Glyceryl Trinitrate
- 4 (Active Comparator): 1.8mg Glyceryl Trinitrate topically to 2 adjacent fingers on non-dominant hand one time
  Interventions: Drug: Glyceryl Trinitrate
- 5 (Active Comparator): 2.4 mg Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand one time
  Interventions: Drug: Glyceryl Trinitrate

INTERVENTIONS:
Drug: placebo cream — placebo cream applied to 2 adjacent fingers of non-dominant hand one time
  Arms: 1.
Drug: Glyceryl Trinitrate — 0.6mg of Glyceryl Trinitrate applied to 2 adjacent fingers on non-dominant hand one time
  Arms: 2
Drug: Glyceryl Trinitrate — 1.2mg Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand one time
  Arms: 3
Drug: Glyceryl Trinitrate — 1.8mg Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand one time
  Arms: 4
Drug: Glyceryl Trinitrate — 2.4 mg Glyceryl Trinitrate topically to 2 adjacent fingers of non-dominant hand one time
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the blood flow response to topical Glyceryl Trinitrate when applied to the skin of patient's fingers with Raynaud's Phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged between 18 and 50 inclusive
* Subject has idiopathic RP (patient may have undifferentiated connective tissue disease with positive ANA) diagnosed for more than two (2) years
* If a female, subject must be non-pregnant and non-lactating
* The subject has provided written informed consent prior to admission to this study

Exclusion Criteria:

* History of clinically relevant medical illnesses (not considering RP) that in the Investigator's opinion may jeopardize subject's safety or interfere with participation in the study, including but not limited to hemoglobinopathy, hemophilia, clinically significant retinal abnormalities, unstable hypertension, liver diseases, chronic pulmonary diseases, significant cardiovascular diseases, diabetes, thyroid diseases, gout, psychiatric or psychological disorders, CNS trauma or active seizure disorders, allergic or immunologically mediated disorders
* History in the past five (5) years of drug or alcohol abuse
* History in the past five (5) years of vascular migraine or other chronic severe headache
* History in the past five (5) years of autonomic neuropathy or postural hypotension
* Unwilling or unable to comply with the restrictions outlined in the protocol
* Current use of smoking cessation treatment, including nicotine patches
* History of drug allergies, anaphylaxis or laryngeal oedema, including allergy to GTN, propylene/ethylene glycol or common moisturizing creams
* Use of any nitrate medication or any phosphodiesterase inhibitor within three (3) days prior to or intended use one (1) day following each dosing with study drug
* Currently treated for hypertension
* Currently receiving treatment for prevention and/or treatment of RP
* Use of any investigational medication within 30 days prior to dosing with study medication or scheduled to receive an investigational drug other than during the course of this study
* Open skin lesions or pathological condition (including, but not limited to, infection) in the area where the study medication is to be applied
* Use of topical corticosteroid to the hand or fingers within 10 days of treatment with study drug
* Withdrawal of consent at any time during the study
* Any condition, which compromises ability to give informed consent or to communicate with the investigator as required for the completion of this study
* Previously enrolled in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Investigate vascular responses to topical Glyceryl Trinitrate versus placebo in patients with Raynaud's using laser Doppler imaging to measure blood flow | 6 visits no less than 10 hours between visits

SECONDARY OUTCOMES:
Evaluate the dose proportionality of the microvascular response to topical Glyceryl Trinitrate | 6 visits no less than 10 hours between visits
Compare the systemic versus topical effect of Glyceryl Trinitrate on vascular response. | 6 visits no less than 10 hours between visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa-Institute for Clinical and Translational Science, Iowa City, Iowa, United States